CLINICAL TRIAL: NCT07402967
Title: Perceptions of Parents and Children on Posterior Restorations in Primary Molars: An Institutional Study
Brief Title: Perceptions of Parents and Children on Posterior Restorations in Primary Molars
Status: Completed | Type: Observational
Sponsor: Universiti Teknologi Mara (Other)
Responsible Party: Principal Investigator, Dr Abdul Rauf Badrul Hisham, Dr, Universiti Teknologi Mara
Other Study IDs: ERC/01/2025 (ERP/4/19) (39)
Record Dates: First submitted 2026-01-20; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Dental Caries; Dental Restorations
Keywords: Perception; Children; Parent; Dental Restoration
MeSH Terms: conditions — Dental Caries | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children: Child aged from 5-12 years old
  Interventions: Other: Questionnaire
- Parent: Parent who had child aged 5-12 years old
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire about their perception on dental restoration for paediatric posterior teeth

SUMMARY:
The research on "Perceptions of Parents and Children on Posterior Restorations in Primary Molars at Universiti Teknologi MARA (UiTM)" gives valuable insights into what influences treatment choices in children's dental care. By understanding the worries and preferences of both parents and children, the study helps dentists better meet their needs, making the experience more comfortable. The findings enhance communication, promote informed decision-making, and ultimately improve patient satisfaction in children's dental care. For parents and children, participating in this research provides a clearer understanding of treatment options, ensures their preferences are considered and creates a more positive dental experience.

This research also helps improve paediatric dentistry overall, promoting family-centered care and guiding future dental practices and policies. The information gathered from this research will benefit individuals, researchers, institutions, and the community by advancing knowledge and informing future practices.

DETAILED DESCRIPTION:
This questionnaire includes demographic questions and one section related to the study. Please be assured that your information will be kept confidential and used exclusively for this research. The questions should take about 10 minutes to complete. Please respond to them to the best of your preference. The outcomes of this study will be critical for assessing parents' and children's perception on tooth fillings at baby molars teeth.

ELIGIBILITY:
Inclusion Criteria:

* Children

  1. Children aged 5-12 years old.
  2. Paediatric patients who attended UiTM undergraduate clinic.
  3. Fit and healthy patient.
  4. Children who understand English or Malay.
* Parents

  1. Parents/guardians who have provided consent to participate in the study.
  2. Parents who understand English or Malay.
  3. Only one parent for each child.

Exclusion Criteria:

Children

1. Children below 5 years old and above 12 years old.
2. Paediatric patients who attended other than UiTM undergraduate clinics.
3. Children with disabilities.
4. Children who do not understand English or Malay.

Parent

1. Parents with children below 5 years old and above 12 years old.
2. Parents/guardians who do not provide consent to participate in the study.
3. Parents who do not understand English or Malay. -

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Who attended UiTM undergraduate clinic.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-16 (Actual)

PRIMARY OUTCOMES:
Parental Preference for Posterior Restorations in Primary Molars | January 2025 until January 2026
  Outcome Measure Description: Assessment of the parents' preferred choice of restoration using the study questionnaire (Domain 3.4: Perception). Parents are presented with 4 images representing different restoration options: Image A (Stainless steel crown), Image B (Amalgam restoration), Image C (Composite restoration), and Image D (Bioflex crown), and asked to select the single option they prefer.
  Unit of Measure: Percentage of participants

SECONDARY OUTCOMES:
Parental Income Level | january 2025 until January 2026
  Outcome Measure Description: Assessment of the parents' socioeconomic status based on self-reported monthly income collected via the sociodemographic section of the study questionnaire.
  Unit of Measure: Malaysian Ringgit (MYR). Grouped into
  Monthly household income :
  Less than RM2499 RM2500 - RM4849 RM4850 - RM 10,959 More than RM11,000
Age of Child | January 2025 until January 2026
  Outcome Measure Description: Assessment of the paediatric patient's age collected via the sociodemographic section of the study questionnaire.
  Unit of Measure: Years (or months, as applicable)
Parental Education Level | January 2025 until January 2026
  Outcome Measure Description: Assessment of the parents' highest level of education attained, collected via the sociodemographic section of the study questionnaire.
  Unit of Measure: Level of education
  No formal education Primary school Secondary school Tertiary school Postgraduate
Gender of Child | January 2025 until January 2026
  Outcome Measure Description: Assessment of the paediatric patient's gender (e.g., male or female) collected via the sociodemographic section of the study questionnaire.
  Unit of Measure: Percentage of participants (e.g., % Male, % Female)

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Teknologi MARA, Sungai Buloh, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided